CLINICAL TRIAL: NCT01366443
Title: Analysis of ROM Plus to Detect Rupture of Membranes
Status: Completed | Type: Observational
Sponsor: Clinical Innovations, LLC (Industry)
Collaborators: Midwestern University (Other); The Reading Hospital and Medical Center (Other); University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: ROM Plus Clinical Study
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Rupture of Amniotic Membranes
Keywords: ROM PLUS; conventional clinical tests of rupture of membranes (ROM); speculum exam; visualization of leakage; pooling of amniotic fluid in the posterior fornix; nitrazine testing; ferning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- women pregnant: Healthy pregnant women between 15 or greater weeks gestation reporting with signs or symptoms of rupture of membranes.
  Interventions: Procedure: Sterile speculum exam; Procedure: ROM Plus Exam; Procedure: Chart Reveiw

INTERVENTIONS:
Procedure: Sterile speculum exam — Sterile vaginal speculum exam to include Nitrazine, ferning and pooling observations
Procedure: ROM Plus Exam — Vaginal swab exam for ROM Plus Test
Procedure: Chart Reveiw — Post delivery blinded chart review by expereienced obstetrician

SUMMARY:
Specific objectives include confirmation: i) that the ROM PLUS consistently and accurately diagnoses rupture of membranes (ROM), ii) that the technique can be understood and applied in clinical practice, and iii) that the ROM PLUS is easier to use than the conventional method.

DETAILED DESCRIPTION:
This study is designed to assess the sensitivity and specificity of ROM PLUS- a rapid, point of care, qualitative immunochromatographic test for the detection (in vitro) of amniotic fluid in cervico-vaginal secretions of women with suspected rupture of membranes (ROM) during pregnancy. The ROM PLUS detects a specific Combo protein present in amniotic fluid of pregnant women in all trimesters of pregnancy. This specific protein combo is unique and found only in amniotic fluid, therefore can be used as a specific marker for the diagnosis of ROM. This biomarker is an isoform of a similar biomarkers called Amni-Sure and ActimProm and was recently approved by the FDA for clinical use. Like these protein markers ( AmniSure or ActimProm) which have been used to diagnose PROM, this particular protein isoform tested for ROM PLUS is in low concentration in other body fluids such as maternal blood, cord blood, urine and semen.

ELIGIBILITY:
Exclusion Criteria:

* Known placental previa
* Active vaginal bleeding

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women between 15 or greater weeks gestation reporting with signs or symptoms of rupture of membranes.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Lee SI, Park JS, Norwitz ER et al. Measurement of placental alpha-microglobulin-1 in cervicovaginal discharge to diagnose rupture of membranes, Obstet Gyencol 2007;109:634-40 Cousins, LM, Smok, P. Lovett, SM, Poeltler, DM. AmniSure Placental Alpha Microglobulin-1 Rapid Immunoassay versus Standard Diagnostic Methods for Detection of Rupture of Membranes. American J. of Perinatology. 2005;Vol.20:1-4. Caughey, AB., Robinson, JN., Norwitz, ER. Contemporary Diagnosis and Management of Preterm Premature Rupture of Membranes. Rev. Obstet. Gynecol. 2008;1(1):11-22.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from July 2010 to May 2011 at three Medical Hospitals, Departments of Obstetric and Gynecology Labor and Delivery Wards.
Pre-assignment Details: No particpants were excluded that matched the particpant enrollment of evaluation for suspicion of rupture of amniotic membranes by standard speculum examination for cervical leaking, pooling, ferning and nitrazine.
Period: Overall Study
Arm/Group | Women Pregnant
Started | 288
Completed | 285
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Under 18 yo | 1

BASELINE CHARACTERISTICS:
Arm/Group | Women Pregnant
Number analyzed (Participants) | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 287
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.26 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 288

OUTCOME MEASURES:

1. Primary Outcome: Pregnant Women Positive and Negative for Membrane Rupture Measured Via Clinical Assessment, Chart Review and ROM Plus
Description: Patients underwent two assessments to determine positive or negative membrane rupture status: (1) Standard clinical assessment using fluid leaking from the cervical os, or two of the following; pooling, positive nitrazine test, or ferning and (2) A new combination immunoassay ROM Plus containing a combination of monoclonal and polyclonal antibodies to Placental Protein 12 (PP12) and Alpha-fetoprotein (AFP). Then, membrane rupture status was determined by chart review for reference based on a post delivery patient chart review by an experienced physician blinded to ROM Plus results.
Time Frame: 1 week
Population: Healthy pregnant women between 15 or greater weeks gestation reporting with signs or symptoms of rupture of membranes who underwent all three assessments.
Measure: Number; unit: participants
Groups:
- Pregnant Women (Clinical Assessment vs. Chart Review): This study was a multi-center prospective observational study performed in patients presenting with signs or symptoms of rupture of amniotic membranes. Initial evaluation included the standard clinical assessment for rupture of membranes. The clinical diagnosis of rupture of membranes was confirmed on review of the medical chart records following delivery.
- Pregnant Women (ROM Plus vs. Chart Review): This study was a multi-center prospective observational study performed in patients presenting with signs or symptoms of rupture of amniotic membranes. Initial evaluation included the new combination immunoassay ROM Plus containing a combination of monoclonal and polyclonal antibodies to Placental Protein 12 (PP12) and Alpha-fetoprotein (AFP). The clinical diagnosis of rupture of membranes was confirmed on review of the medical chart records following delivery.
Arm/Group | Pregnant Women (Clinical Assessment vs. Chart Review) | Pregnant Women (ROM Plus vs. Chart Review)
Number analyzed (Participants) | 285 | 285
participants
  True Negative Membrane Rupture | 95 [0.97 to 1.00] | 88
  True Positive Membrane Rupture | 160 | 187
  False Negative Membrane Rupture | 2 | 9
  False Positive Membrane Rupture | 28 | 1
Statistical Analysis 1: Comparison: Pregnant Women (Clinical Assessment vs. Chart Review); Sensitivity = true positives/(true positives + false negatives); It indicates how likely is the test to detect the presence of a characteristic in someone with the characteristic; Test type: Superiority or Other; Sensitivity = 0.85, 95% CI 2-sided [0.79 to 0.89] — The calculation for the Wilson CI is computed using the cii (confidence interval immediate) command in Stata version 11.2, with the "Wilson" option
Statistical Analysis 2: Comparison: Pregnant Women (Clinical Assessment vs. Chart Review); Specificity = true negatives/(false positives + true negatives); It indicates how likely the test is to detect the absence of a characteristic in someone without the characteristic; Test type: Superiority or Other; Specificity = 0.98, 95% CI 2-sided [0.93 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pregnant Women (Clinical Assessment vs. Chart Review); Positive Predictive Value = true positives/(true positives + false positives); It indicates how likely it is that someone with a positive test result will actually have the characteristic; Test type: Superiority or Other; Positive Predictive Value = 0.99, 95% CI 2-sided [0.96 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Pregnant Women (Clinical Assessment vs. Chart Review); Negative Predictive Value = true negatives/(true negatives + false negatives); It indicates how likely it is that someone with a negative test result will actually not have the characteristic; Test type: Superiority or Other; Negative Predictive Value = 0.77, 95% CI 2-sided [0.69 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Pregnant Women (ROM Plus vs. Chart Review); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Sensitivity = 0.99, 95% CI 2-sided [0.97 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Pregnant Women (ROM Plus vs. Chart Review); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Specificity = 0.91, 95% CI 2-sided [0.83 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Pregnant Women (ROM Plus vs. Chart Review); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Positive Predictive Value = 0.95, 95% CI 2-sided [0.90 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Pregnant Women (ROM Plus vs. Chart Review); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Negative Predictive Value = 0.99, 95% CI 2-sided [0.94 to 1.00] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Women Pregnant
Serious Adverse Events (participants affected / at risk) | 0/288
Other Adverse Events (participants affected / at risk) | 0/288

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No